CLINICAL TRIAL: NCT02168049
Title: Heart and Lung Function Monitoring System Evaluation
Brief Title: Heart and Lung Function Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ICR14-000670
Record Dates: First submitted 2014-06-11; First posted 2014-06-20 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Heart Diseases; Lung Diseases
Keywords: cardiac, respiratory, monitoring
MeSH Terms: conditions — Heart Diseases; Lung Diseases | interventions — Echocardiography; Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Heart and Lung Function Monitioring (Experimental)
  Interventions: Device: Integrated CardioRespiratory System; Device: Transthoracic Echocardiography (TTE); Device: Electrocardiography

INTERVENTIONS:
Device: Integrated CardioRespiratory System — Participants will be asked to wear a non-invasive band on their upper abdomen while laying down. This band includes acoustic sensors. A remote monitoring device will continuously monitor and record heart rate and lung volumes and function.
Device: Transthoracic Echocardiography (TTE) — Participants will undergo a TTE examination. During the TTE, a technician obtains views of the heart by moving a small instrument called a transducer to different locations on the chest or abdominal wall.
Device: Electrocardiography — Participants will also have ECG monitoring as part of the TTE exam, which records the electrical activity of the heart using electrodes placed on the body.
  Other Names: ECG

SUMMARY:
The investigator goal is to test a new device to see if it can provide continuous and simultaneous monitoring of heart and lung function.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and guide progress in the development of a new instrument that may provide continuous, integrated monitoring of heart and lung function.

ELIGIBILITY:
Inclusion Criteria:

* Adult's ≥ 18 years old

Exclusion Criteria:

* Wounds, surgical incisions at the site of sensor placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Acoustic heart sound electronic data | 60 minutes during system trial
  Heart and lung function monitoring

SECONDARY OUTCOMES:
Standard echocardiography parameters | 60 minutes during examination simultaneous with system trial
  Transthoracic Echocardiography (TTE)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Howard-Quijano, M.D., M.S., Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No